CLINICAL TRIAL: NCT01866592
Title: Vascular Inflammation in Psoriasis - Extension Study
Acronym: VIP-E
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 817552
Record Dates: First submitted 2013-05-16; First posted 2013-05-31 (Estimated); Results first posted 2018-05-22 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Psoriasis; Cardiovascular Disease
Keywords: Psoriasis; Cardiovascular Disease; Vascular Inflammation; Lipid Biomarkers; Metabolic biomarkers; FDG-PET/CT
MeSH Terms: conditions — Psoriasis; Cardiovascular Diseases | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single-Arm, open-label extension trial (Other): Single-arm, open label extension trial to continue treatment with Humira (Adalimumab) subcutaneous injection 80mg initial dose followed by 40mg maintenance dose every other week for up to 52 weeks.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Study participants will receive the FDA-approved dosing schedule for Adalimumab (Humira): an initial dose of 80mg followed by a 40mg maintenance dose every other week up to 52 weeks.
  Other Names: Humira

SUMMARY:
VIP-E is a one-arm, open-label, 40-52 week extension study to continue or cross over subjects of the VIP study (# 814278) to active drug (adalimumab) to determine if there is sustained improvement in vascular inflammation, lipid metabolism, and inflammatory markers. VIP-E extends VIP study procedures for 40-52 weeks including questionnaires, physical exams, blood and urine samples, lab tests, one additional FDG-PET/CT scan, and adalimumab injections following FDA-approved psoriasis treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years of age and older.
2. Subject completed the VIP Study
3. Subject willing and able to avoid prolonged exposure of skin affected by psoriasis to natural or sunlight or tanning beds during the course of the study
4. Subject is willing and able to avoid topical or systemic prescription treatments for psoriasis besides adalimumab during the course of the study
5. Women are eligible to participate in the study if they meet one of the following criteria:

   1. Women of childbearing potential must undergo pregnancy testing during the baseline visit and agree to use one of the following methods of contraception throughout the 13-month study:

      * Oral contraceptives;
      * Transdermal contraceptives
      * Injectable or implantable methods
      * Intrauterine devices
      * Barrier methods (for example but not limited to a diaphragm with spermicide, condom with spermicide); or
      * Vasectomized partner
      * Subjects using oral or parental forms of contraceptives must have been using those methods of birth control for at least three months prior to the baseline visit.
   2. Women who have undergone tubal ligation
   3. Women who are postmenopausal (for at least one year), sterile, or hysterectomized are eligible to participate
   4. Women who agree to be sexually abstinent, defined as total abstinence from sexual intercourse, as a form of contraception are eligible to participate in the study.
6. Subject is judged to be in good general health as determined by the Principal Investigator based upon the results of medical history, laboratory profile, and physical examination.
7. Able and willing to give written informed consent and to comply with requirements of this study protocol.

Exclusion Criteria:

1. Previous adverse event following exposure to a TNF-alpha antagonist that led to discontinuation of the TNF inhibitor and contraindicates future treatment.
2. Previous lack of response to a TNF-alpha antagonist led to discontinuation.
3. Diagnosis of erythrodermic psoriasis, generalized pustular psoriasis, or medication-induced or medication-exacerbated psoriasis.
4. Diagnosis of other active skin diseases or skin infections (bacterial, fungal, or viral) that may interfere with evaluation of psoriasis.
5. Subject is taking or requires oral or injectable corticosteroids during the study. Inhaled corticosteroids for stable medical conditions are allowed.
6. Poorly controlled medical condition, such as unstable ischemic heart disease, congestive heart failure, recent cerebrovascular accidents, psychiatric disease requiring frequent hospitalization, and any other condition, which, in the opinion of the Investigator, would put the subject at risk by participation in the study.
7. History of diabetes mellitus, type 1 or type 2 (patients with type 2 diabetes may be enrolled if the duration of diabetes is <10 years and HbA1c is <7.0%)
8. Uncontrolled hypertension, with measured systolic blood pressure >180 mmHg or diastolic blood pressure >90 mmHg
9. History of demyelinating diseases or lupus.
10. Subject has infection or risk factors for severe infections, for example:

    * Known history of HIV, hepatitis B or C, or other severe, recurrent, or persistent infections;
    * Excessive immunosuppression or other factors associated with it, including human immunodeficiency virus infection;
    * Active tuberculosis (TB) disease;
    * Evidence of latent TB infection demonstrated by Purified Protein Derivative (PPD) ≥ 5 mm of induration or positive Quantiferon-GOLD results as determined within 6 months of the baseline visit for VIP-E; except if prophylactic treatment for TB, as recommended by local guidelines, is initiated prior to administration of study drug or if there is documentation that the subject has received prophylactic treatment for TB previously.
    * Any other significant infection requiring hospitalization or intravenous (IV) antibiotics in the month prior to Baseline;
    * Infection requiring treatment with oral or parenteral antibiotics within 14 days prior to Baseline;
    * Subject will require a live vaccination during study participation including up to 30 days after the last dose of study drug.
11. Subject has history of hematological or solid malignancy within the past five years other than successfully treated basal cell carcinoma, non-metastatic cutaneous squamous cell carcinoma or cervical carcinoma in situ.
12. Female subject who is pregnant or breast-feeding or considering becoming pregnant during the study.
13. Clinic laboratory analyses showing any of the following abnormal results:

    * Hemoglobin (Hgb) < 10 g/dL in females or <12 g/dL in males;
    * White blood cell (WBC) count <2.5 x 109/L

      * Subject can be included if WBC count is <2.5 x x 109/L and absolute neutrophil count (ANC) is >1000 cells / mm3.
    * WBC count > 15 x 109/L;
    * Platelet count < 100 x 109/L;
    * Serum aspartate transaminase (AST) or alanine transaminase (ALT) >2.5 upper limits of normal (ULN);
    * Serum total bilirubin ≥2 mg/dL (≥26 µmol/L)
14. Recent history of substance abuse or psychiatric illness that could preclude compliance with the protocol.
15. If subject is on cholesterol-lowering medication (e.g. statin), dose and form of medication must be stable for 90 days prior to baseline and remain stable throughout the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-04; Primary Completion 2016-08-08 (Actual); Study Completion 2016-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel M Gelfand, MD MSCE, Principal Investigator — University of Pennsylvania
Locations (9):
- United States (9):
  - University of California, Davis Health System, Sacramento, California
  - University of Colorado, Denver, Colorado
  - National Heart, Lung, and Blood Institute, Bethesda, Maryland
  - Buffalo Medical Group, Buffalo, New York
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Menter Dermatology Research Institute, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Mehta NN, Shin DB, Joshi AA, Dey AK, Armstrong AW, Duffin KC, Fuxench ZC, Harrington CL, Hubbard RA, Kalb RE, Menter A, Rader DJ, Reilly MP, Simpson EL, Takeshita J, Torigian DA, Werner TJ, Troxel AB, Tyring SK, Vanderbeek SB, Van Voorhees AS, Playford MP, Ahlman MA, Alavi A, Gelfand JM. Effect of 2 Psoriasis Treatments on Vascular Inflammation and Novel Inflammatory Cardiovascular Biomarkers: A Randomized Placebo-Controlled Trial. Circ Cardiovasc Imaging. 2018 Jun;11(6):e007394. doi: 10.1161/CIRCIMAGING.117.007394. PMID 29776990

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single-Arm, Open-label Extension Trial
Started | 81
Completed | 58
Not Completed | 23

BASELINE CHARACTERISTICS:
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8642 (14.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 63
  More than one race | 0
  Unknown or Not Reported | 4
Psoriasis Duration [Mean (Standard Deviation); unit: years] — Population: Two participants did not respond to question, missing data.
  years
    number analyzed (Participants) | 79
    (all) | 16.27 (13.78)
Psoriatic Arthritis [Count of Participants; unit: Participants] — Population: Two participants did not respond to question, missing data.
  Participants
    number analyzed (Participants) | 79
    (all) | 9
History of Cardiovascular Disease [Count of Participants; unit: Participants] | 6
Diabetes [Count of Participants; unit: Participants] | 3
History of Hypertension [Count of Participants; unit: Participants] | 14
History of Hyperlipidemia [Count of Participants; unit: Participants] | 11
History of Statin Use [Count of Participants; unit: Participants] | 7
10 year Framingham Risk [Mean (Standard Deviation); unit: percentage] — Absolute risk of developing a first cardiovascular disease (CVD) event (coronary death, myocardial infarction, coronary insufficiency, angina, ischemic stroke, hemorrhagic stroke, transient ischemic attack, peripheral artery disease, heart failure) within 10 years. The units are in 10-year risk percentage.
  percentage | 7.44 (8.3)
Body Surface Area [Mean (Standard Deviation); unit: kg/m^2] | 24.37 (14.65)
PASI (Psoriasis Area and Severity Index) [Mean (Standard Deviation); unit: units on a scale] — PASI combines the assessment of the severity of lesions and the area affected into a single score in the range of 0 (no disease) to 72 (maximal disease).
  units on a scale | 19.12 (7.41)
PGA (Physician's Global Assessment) [Mean (Standard Deviation); unit: units on a scale] — The PGA is an average assessment of all psoriatic lesions based on erythema, scale, and induration with scores ranging from 0 (no disease) to 5 (maximal disease).
  units on a scale | 3.25 (.59)
DLQI (Dermatology Quality of Life Index) [Mean (Standard Deviation); unit: units on a scale] — The DLQI is calculated by summing the score of 10 questions regarding impact of skin condition on daily life resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
  units on a scale | 15.02 (6.52)
History of Phototherapy [Count of Participants; unit: Participants] — Population: Data was collected after last follow up visit, only 50 of 81 participants responded.
  Participants
    number analyzed (Participants) | 50
    (all) | 23
History of Oral Systemics [Count of Participants; unit: Participants] — Population: Data was collected after last follow up visit, only 50 of 81 participants responded.
  Participants
    number analyzed (Participants) | 50
    (all) | 28
History of Biologics [Count of Participants; unit: Participants] — Population: Data was collected after last follow up visit, only 50 of 81 participants responded.
  Participants
    number analyzed (Participants) | 50
    (all) | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Vascular Inflammation
Description: Change in total vascular inflammation of five aortic segments as assessed on FDG-PET/CT between week 52 of the adalimumab treatment period and baseline scans (prior to randomization in the VIP Trial). The arterial uptake of FDG is measured by the standardized uptake value (SUV) max divided by the venous SUIV mean yielding a target to background ration (TBR). If subjects were randomized to adalimumab in the VIP Trial, the time frame is a total of 52 weeks (continuation group). If subjects were randomized to placebo or phototherapy in the VIP Trial, additional 12 weeks added to the time frame for a total of 64 weeks (crossover group).
Time Frame: 52 weeks (continuation group) or 64 weeks (crossover group)
Measure: Number (95% Confidence Interval); unit: percentage change
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
percentage change | -3.8 [-6.4 to -1.19]

2. Primary Outcome: Change in Vascular Inflammation
Description: Change in total vascular inflammation of five aortic segments as assessed on FDG-PET/CT between week 52 of the adalimumab treatment period and start of adalimumab.The arterial uptake of FDG is measured by the standardized uptake value (SUV) max divided by the venous SUIV mean yielding a target to background ration (TBR).
Time Frame: 52 weeks of adalimumab treatment
Measure: Number (95% Confidence Interval); unit: percentage change
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
percentage change | 0.02 [-2.85 to 2.90]

3. Primary Outcome: Change in Cardiometabolic Biomarker - Total Cholesterol
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - Total Cholesterol. If subjects were randomized to adalimumab in the VIP Trial, the time frame is a total of 52 weeks (continuation group). If subjects were randomized to placebo or phototherapy in the VIP Trial, additional 12 weeks added to the time frame for a total of 64 weeks (crossover group).
Time Frame: 52 weeks (continuation group) or 64 weeks (crossover group)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
mg/dL | 3.164 (4.216)

4. Primary Outcome: Change in Cardiometabolic Biomarker - Cholesterol Efflux
Description: The ability to promote cholesterol efflux from macrophages is a classic function of HDL that is thought to be an important mechanism by which HDL protects against atherosclerosis. HDL cholesterol efflux capacity assays are performed based on published methods using J774 cells derived from a murine macrophage cell line (Mehta NN Atherosclerosis 2012). Efflux is calculated as a unitless measure by using the following formula: [(µCi of 3H-cholesterol in media containing apoB-depleted subject plasma - µCi of 3H-cholesterol in plasma-free media) / (µCi of 3H-cholesterol in media containing apoB-depleted pooled control plasma-µCi of 3H-cholesterol in pooled control plasma-free media)].
  If subjects were randomized to adalimumab in the VIP Trial, the time frame is a total of 52 weeks (continuation group). If subjects were randomized to placebo or phototherapy in the VIP Trial, additional 12 weeks added to the time frame for a total of 64 weeks (crossover group).
Time Frame: 52 weeks (continuation group) or 64 weeks (crossover group)
Measure: Mean (Standard Error); unit: no units
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
no units | -0.217 (0.032)

5. Primary Outcome: Change in Cardiometabolic Biomarker - Low-density Lipoprotein Particle
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - Low-density lipoprotein particle If subjects were randomized to adalimumab in the VIP Trial, the time frame is a total of 52 weeks (continuation group). If subjects were randomized to placebo or phototherapy in the VIP Trial, additional 12 weeks added to the time frame for a total of 64 weeks (crossover group).
Time Frame: 52 weeks (continuation group) or 64 weeks (crossover group)
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
nmol/L | 22.537 (44.283)

6. Primary Outcome: Change in Cardiometabolic Biomarker - High-density Lipoprotein Particle
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - High-density lipoprotein particle If subjects were randomized to adalimumab in the VIP Trial, the time frame is a total of 52 weeks (continuation group). If subjects were randomized to placebo or phototherapy in the VIP Trial, additional 12 weeks added to the time frame for a total of 64 weeks (crossover group).
Time Frame: 52 weeks (continuation group) or 64 weeks (crossover group)
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
nmol/L | -2.984 (.786)

7. Primary Outcome: Change in Cardiometabolic Biomarker - Log Insulin
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - Log Insulin If subjects were randomized to adalimumab in the VIP Trial, the time frame is a total of 52 weeks (continuation group). If subjects were randomized to placebo or phototherapy in the VIP Trial, additional 12 weeks added to the time frame for a total of 64 weeks (crossover group).
Time Frame: 52 weeks (continuation group) or 64 weeks (crossover group)
Measure: Mean (Standard Error); unit: log(pg/mL)
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
log(pg/mL) | .118 (.136)

8. Primary Outcome: Change in Cardiometabolic Biomarker - Log Adiponectin
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - Log Adiponectin If subjects were randomized to adalimumab in the VIP Trial, the time frame is a total of 52 weeks (continuation group). If subjects were randomized to placebo or phototherapy in the VIP Trial, additional 12 weeks added to the time frame for a total of 64 weeks (crossover group).
Time Frame: 52 weeks (continuation group) or 64 weeks (crossover group)
Measure: Mean (Standard Error); unit: log(ug/mL)
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
log(ug/mL) | -.074 (.068)

9. Primary Outcome: Change in Cardiometabolic Biomarker - Log Leptin
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - Log Leptin If subjects were randomized to adalimumab in the VIP Trial, the time frame is a total of 52 weeks (continuation group). If subjects were randomized to placebo or phototherapy in the VIP Trial, additional 12 weeks added to the time frame for a total of 64 weeks (crossover group).
Time Frame: 52 weeks (continuation group) or 64 weeks (crossover group)
Measure: Mean (Standard Error); unit: log(pg/mL)
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
log(pg/mL) | .048 (.195)

10. Primary Outcome: Change in Cardiometabolic Biomarker - Log C-reactive Protein
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - Log C-reactive protein If subjects were randomized to adalimumab in the VIP Trial, the time frame is a total of 52 weeks (continuation group). If subjects were randomized to placebo or phototherapy in the VIP Trial, additional 12 weeks added to the time frame for a total of 64 weeks (crossover group).
Time Frame: 52 weeks (continuation group) or 64 weeks (crossover group)
Measure: Mean (Standard Error); unit: log(pg/mL)
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
log(pg/mL) | -.815 (.192)

11. Primary Outcome: Change in Cardiometabolic Biomarker - Log Tumor Necrosis Factor-Alpha
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - Log Tumor Necrosis Factor-Alpha If subjects were randomized to adalimumab in the VIP Trial, the time frame is a total of 52 weeks (continuation group). If subjects were randomized to placebo or phototherapy in the VIP Trial, additional 12 weeks added to the time frame for a total of 64 weeks (crossover group).
Time Frame: 52 weeks (continuation group) or 64 weeks (crossover group)
Measure: Mean (Standard Error); unit: log(pg/mL)
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
log(pg/mL) | -.275 (.131)

12. Primary Outcome: Change in Cardiometabolic Biomarker - Log Interleukin 6
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - Log Interleukin 6 If subjects were randomized to adalimumab in the VIP Trial, the time frame is a total of 52 weeks (continuation group). If subjects were randomized to placebo or phototherapy in the VIP Trial, additional 12 weeks added to the time frame for a total of 64 weeks (crossover group).
Time Frame: 52 weeks (continuation group) or 64 weeks (crossover group)
Measure: Mean (Standard Error); unit: log(pg/mL)
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
log(pg/mL) | 1.054 (.243)

13. Primary Outcome: Change in Cardiometabolic Biomarker - GlycA
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - GlycA If subjects were randomized to adalimumab in the VIP Trial, the time frame is a total of 52 weeks (continuation group). If subjects were randomized to placebo or phototherapy in the VIP Trial, additional 12 weeks added to the time frame for a total of 64 weeks (crossover group).
Time Frame: 52 weeks (continuation group) or 64 weeks (crossover group)
Measure: Mean (Standard Error); unit: log(pg/mL)
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
log(pg/mL) | -29.559 (7.749)

14. Primary Outcome: Change in Cardiometabolic Biomarkers: - Total Cholesterol
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and the start of adalimumab - Total Cholesterol
Time Frame: 52 weeks of adalimumab treatment
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
mg/dL | 1.194 (3.746)

15. Primary Outcome: Change in Cardiometabolic Biomarker - Cholesterol Efflux
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - Cholesterol Efflux
Time Frame: 52 weeks of adalimumab treatment
Measure: Mean (Standard Error); unit: no units
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
no units | -.225 (.030)

16. Primary Outcome: Change in Cardiometabolic Biomarker - Low-density Lipoprotein Particle
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - Low-density lipoprotein particle
Time Frame: 52 weeks of adalimumab treatment
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
nmol/L | 23.313 (42.860)

17. Primary Outcome: Change in Cardiometabolic Biomarker - High-density Lipoprotein Particle
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - High-density lipoprotein particle
Time Frame: 52 weeks of adalimumab treatment
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
umol/L | -2.630 (.778)

18. Primary Outcome: Change in Cardiometabolic Biomarker - Log Insulin
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - Log Insulin
Time Frame: 52 weeks of adalimumab treatment
Measure: Mean (Standard Error); unit: log(pg/mL)
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
log(pg/mL) | .188 (.134)

19. Primary Outcome: Change in Cardiometabolic Biomarker - Log Adiponectin
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - Log Adiponectin
Time Frame: 52 weeks of adalimumab treatment
Measure: Mean (Standard Error); unit: log(ug/mL)
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
log(ug/mL) | -.055 (.067)

20. Primary Outcome: Change in Cardiometabolic Biomarker - Log Leptin
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - Log Leptin
Time Frame: 52 weeks of adalimumab treatment
Measure: Mean (Standard Error); unit: log(pg/mL)
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
log(pg/mL) | .077 (.201)

21. Primary Outcome: Change in Cardiometabolic Biomarker - Log C-reactive Protein
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - Log C-reactive protein
Time Frame: 52 weeks of adalimumab treatment
Measure: Mean (Standard Error); unit: log(pg/mL)
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
log(pg/mL) | -.615 (.189)

22. Primary Outcome: Change in Cardiometabolic Biomarker - Log Tumor Necrosis Factor-Alpha
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - Log Tumor Necrosis Factor-Alpha
Time Frame: 52 weeks of adalimumab treatment
Measure: Mean (Standard Error); unit: log(pg/mL)
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
log(pg/mL) | -.197 (.132)

23. Primary Outcome: Change in Cardiometabolic Biomarker - Log Interleukin 6
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - Log Interleukin 6
Time Frame: 52 weeks of adalimumab treatment
Measure: Mean (Standard Error); unit: log(pg/mL)
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
log(pg/mL) | 1.309 (.232)

24. Primary Outcome: Change in Cardiometabolic Biomarker - GlycA
Description: Change in metabolic, lipid, and inflammatory biomarker levels between week 52 of the adalimumab treatment period and baseline assessments from the VIP trial - GlycA
Time Frame: 52 weeks of adalimumab treatment
Measure: Mean (Standard Error); unit: log(pg/mL)
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
log(pg/mL) | -17.454 (7.394)

25. Secondary Outcome: Psoriasis Activity (PASI and PGA)
Description: Change in psoriasis activity will be assessed using the following standardized measurement tools for psoriasis: Psoriasis Area and Severity Index (PASI) and Physician's Global Assessment (PGA). PASI combines the assessment of the severity of lesions and the area affected into a single score with range 0 (no disease) to 72 maximal disease. The PGA is an average assessment of all psoriatic lesions based on erythema, scale, and induration with score range 0 (no disease/clear) to 5 (maximal disease).
  If subjects were randomized to adalimumab in the VIP Trial, the time frame is a total of 52 weeks (continuation group). If subjects were randomized to placebo or phototherapy in the VIP Trial, additional 12 weeks added to the time frame for a total of 64 weeks (crossover group).
Time Frame: 52 weeks (continuation group) or 64 weeks (crossover group)
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
Participants
  PASI 75 | 40
  PGA Clear/Almost Clear | 35

26. Secondary Outcome: Safety/Adverse Events
Description: Safety will be assessed by evaluating all subject reported adverse events through the duration of the study.
Time Frame: Baseline - Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 81
Participants
  upper respiratory infection | 11
  musculoskeletal pain | 6

27. Secondary Outcome: Change in Patient-Reported Quality of Life Outcomes-EuroQol EQ-5D
Description: EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ-5D consists of a descriptive system and the EQ VAS. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression on a scale ranging from 1 (no health state problem) to 3 (extreme health state problems). The EQ VAS records the patient's self-rated health on a vertical visual analogue scale ranging from 0, worst health state, to 100, best health state. A scoring function is used to assign a value (i.e., EQ-5D™ index score) to self-reported health states from a set of population-based preference weights. For the U.S. general population, the possible EQ-5D index scores range from -0.11 to 1.0 where 0.0 = death and 1.0 = perfect health.
Time Frame: 52 weeks (continuation group) or 64 weeks (crossover group)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
units on a scale | .09 [.04 to .14]

28. Secondary Outcome: Change in Patient-Reported Quality of Life Outcomes - Dermatology Life Quality Index (DLQI)
Description: The DLQI is calculated by summing the score of 10 questions regarding impact of skin condition on daily life resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
  If subjects were randomized to adalimumab in the VIP Trial, the time frame is a total of 52 weeks (continuation group). If subjects were randomized to placebo or phototherapy in the VIP Trial, additional 12 weeks added to the time frame for a total of 64 weeks (crossover group).
Time Frame: 52 weeks (continuation group) or 64 weeks (crossover group)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
units on a scale | -9.37 [-11.14 to -7.61]

29. Secondary Outcome: Change in Patient-Reported Quality of Life Outcomes - MEDFICTS Dietary Assessment
Description: Patient reported dietary outcomes will be assessed using MEDFICTS (Meats, Eggs, Dairy, Fried foods, fat In baked goods, Convenience foods, fats added at the Table, and Snacks), a brief dietary assessment instrument. This assessment looks at eight different categories of foods and assigns points by type of food and serving size ranging from 0 points (do not consume that food group) to 21 points (consume food group, largest serving size). Your final score is the total of all points for all food categories.
  If subjects were randomized to adalimumab in the VIP Trial, the time frame is a total of 52 weeks (continuation group). If subjects were randomized to placebo or phototherapy in the VIP Trial, additional 12 weeks added to the time frame for a total of 64 weeks (crossover group).
Time Frame: 52 weeks (continuation group) or 64 weeks (crossover group)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
units on a scale | -10.9 [-16.7 to -5.12]

30. Secondary Outcome: Change in Patient-Reported Quality of Life Outcomes - International Physical Activity Questionnaire (IPAQ)
Description: IPAQ is an instrument designed primarily for population surveillance of physical activity among adults with activity measured in metabolic equivalent (MET)-minutes per week.
  Per Office of Disease Prevention and Health Promotion's Physical Activity Guidelines:
  A range of 500 to 1,000 MET-minutes of activity per week provides substantial [health] benefit, and amounts of activity above this range have even more benefit. Amounts of activity below this range also have some benefit. The dose-response relationship continues even within the range of 500 to 1,000 MET-minutes, in that the health benefits of 1,000 MET-minutes per week are greater than those of 500 MET-minutes per week.
  If subjects were randomized to adalimumab in the VIP Trial, the time frame is a total of 52 weeks (continuation group). If subjects were randomized to placebo or phototherapy in the VIP Trial, additional 12 weeks added to the time frame for a total of 64 weeks (crossover group).
Time Frame: 52 weeks (continuation group) or 64 weeks (crossover group)
Measure: Mean (95% Confidence Interval); unit: MET-minutes per week
Arm/Group | Single-Arm, Open-label Extension Trial
Number analyzed (Participants) | 67
MET-minutes per week | 459 [-1233 to 2150]

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Single-Arm, Open-label Extension Trial
Serious Adverse Events (participants affected / at risk) | 1/81
Other Adverse Events (participants affected / at risk) | 16/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-Arm, Open-label Extension Trial (N=81)
syncope (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-Arm, Open-label Extension Trial (N=81)
upper respiratory infection (Infections and infestations) | 11 (11)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes